CLINICAL TRIAL: NCT05305911
Title: Sodium Glucose Co-Transporter 2 (SGLT2) Inhibition Improves Left Ventricular Function and Reduces Adverse Left-Ventricular Remodeling in High-Risk Patients with Microvascular Obstruction (MVO) Following ST-elevation Myocardial Infarction (STEMI).
Brief Title: Sodium Glucose Co-Transporter 2 (SGLT2) and STEMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1852152
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Heart Attack; Enlarged Heart
Keywords: Dapagliflozin; Sodium Glucose Co-Transporter 2
MeSH Terms: conditions — Myocardial Infarction; Cardiomegaly | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Treatment will be blinded to the participant and investigator. Assignment of treatment arm will be managed by Abbott Northwestern Heart Hospital pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Active Comparator): Treatment group will receive SGLT2 inhibitor in addition to standard heart attack medications for the duration of hospitalization and 6-month duration of the study.
  Interventions: Drug: SGLT-2 inhibitors
- Placebo Group (Placebo Comparator): Placebo Group will receive placebo in addition to standard heart attack medications for the duration of hospitalization and 6-month duration of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGLT-2 inhibitors — SGLT2 inhibitor once daily for six months
  Arms: Treatment Group
Drug: Placebo — Placebo once daily for six months
  Arms: Placebo Group

SUMMARY:
The purpose of the research is to determine whether a class of medication called SGLT2 inhibitor will improve the heart's function and reduce its enlargement after a heart attack. Participation in this study will involve taking this class of medication (or a placebo) once daily for six months, one cardiac magnetic resonance imaging (MRI) test during your initial hospitalization, follow-up phone calls at 1 and 3 months, and one cardiac MRI and clinic visit at six months. This is a single center study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with their first STEMI (>18 years) who underwent successful primary PCI and able to give informed consent
* At least mild LV dysfunction (LVEF < 50%) on echocardiogram, cMRI or Left Ventriculargram following PCI
* Infarct size that is > 10% of LV mass
* The presence of MVO that is > 10% of infarct size

Exclusion Criteria:

* Contraindication to cardiac MRI
* Life expectancy < 1 year
* Previous CABG or Valve Surgery
* Previous STEMI
* Pregnant or planning to become pregnant or lactating women
* Cardiogenic shock (not resolved)
* Atrial fibrillation or recurrent sustained ventricular arrhythmias (excluding PVCs)
* GFR<30 ml/min/1.73m2 or end-stage renal disease on dialysis
* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Type I or II diabetes with insulin use
* Prior intolerance of SGLT2 inhibitors
* Current use of SGLT2 inhibitors (randomized patients only)
* Contraindications to gadolinium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in LVESVI | 6 Months
  Change in LVESVI at 6 months as measured by MRI.
Change in LVEDVI | 6 Months
  Change in LVEDVI at 6 months as measured by MRI.

SECONDARY OUTCOMES:
Change in LV mass | 6 months
  Change in LV mass at 6 months as measured by cMRI
Change in LVEF | 6 months
  Change in LVEF at 6 months as measured by cMRI
MACE rates - including hospitalization for CHF, repeat revascularization, MI and death and ICD implantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jay Traverse, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No